CLINICAL TRIAL: NCT00132535
Title: Influence of HIV Infection on the Effectiveness of Malaria Prevention During Pregnancy, With Emphasis on the Effect of Chloroquine on HIV Viral Load Among Pregnant Women in Uganda
Brief Title: Influence of Chloroquine on HIV Viral Load Among Pregnant Women in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: DBL -Institute for Health Research and Development (Other); Uganda AIDS Commission (Unknown)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: MV-714-624-03-0001
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria in Pregnancy; HIV Infections
Keywords: Malaria in pregnancy; IPT; Sulphadoxine-pyrimethamine; Chloroquine; HIV; Viral load; birth weight; anaemia
MeSH Terms: conditions — HIV Infections; Birth Weight; Anemia | interventions — Chloroquine

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine intermittent preventive treatment
Drug: chloroquine

SUMMARY:
There is conflicting evidence regarding the influence of HIV infection on the success of malaria prevention in pregnancy and effect on pregnancy outcome. The purpose of the proposed study is to assess the impact of HIV infection on the effectiveness of malaria prevention during pregnancy. This will be carried out by comparing two intermittent preventive treatments (IPTs) with sulfadoxine/pyrimethamine (SP) plus 300 mg weekly chloroquine with two doses IPT plus a weekly chloroquine placebo. The emphasis will be on assessing the effect of chloroquine on HIV viral load and malaria morbidity and foetal outcome.

The study will be a randomised double-blind placebo-controlled trial with two arms, involving pregnant women attending antenatal classes (ANCs) at health units, enrolled early in their second trimester at 3 health units of the Mbarara district and Kampala. All pregnant women presenting for antenatal care, irrespective of parity, who consent to participate will be enrolled. Women with severe systemic disease or symptoms of AIDS will be excluded from the study data analysis.

Women will be screened for HIV status and their HIV viral loads will be measured at enrolment. Parasitaemia will be assessed at enrolment; at the beginning of the third trimester; and at delivery. Haemoglobin will be measured at the same time points.

The main outcome variables to be assessed will be maternal peripheral parasitaemia; placental parasitaemia; maternal clinical malaria; congenital parasitaemia; and maternal and neonatal haemoglobin, birth weight and viral load at enrolment and before nevirapine administration to the HIV positive mothers at birth.

Anthropological pre-studies to assess the quality of ANC services and healthcare seeking practices of pregnant women in the study area will be carried out. Focus group discussions (FGD) with pregnant women and mothers of neonates; in-depth interviews with relevant health workers; and illness narratives from pregnant women will be used to collect data. The anthropological study results will assist in appropriately planning for the trial to enhance compliance to the intervention.

The data collection is planned to commence in August 2003 and is expected to end in October 2005. Twelve months will be spent on the write-up phase.

DETAILED DESCRIPTION:
General Objective:

* To contribute to the improvement of quality and effectiveness of maternity care services by assessing the impact of HIV infection on the effectiveness of IPT with SP and comparing it with SP plus weekly chloroquine (CQ) to assess the possible anti-retroviral effect of chloroquine.

Specific Objectives:

* To assess the impact of IPT with SP plus placebo CQ or SP plus prophylaxis with CQ on peripheral and placental parasitaemia among HIV sero-positive as compared to HIV sero-negative pregnant women.
* To assess the effect of HIV infection on maternal malaria-related morbidity among pregnant HIV sero-positive women compared to pregnant HIV sero-negative women treated with SP plus placebo CQ or SP plus weekly CQ prophylaxis.
* To describe the effect of HIV infection on birth weight and congenital parasitaemia among babies born to women given IPT with SP as compared to women given SP plus CQ prophylaxis during pregnancy.
* To assess anti-HIV effects of CQ among HIV positive pregnant women by measuring HIV viral load at enrolment and before delivery.

Subsidiary Objectives:

* To explore mothers' and health care providers' perceptions of the quality of maternity services in the study communities.
* To explore fever prevention and management options used by pregnant women in the study communities.
* To explore pregnant women's perceptions of malaria prevention during pregnancy in the era of HIV/AIDS.

Material and Methods:

All pregnant women who present at a gestational age of 14- 24 weeks who will give verbal informed consent will be enrolled in the study from the 2 health units in Mbarara District and a hospital in Kampala. These areas are reported to be highly endemic for malaria. The district has a high prevalence of HIV (10.6%) among antenatal attendants. The main ethnic groups in the area are Banyankore with few migrant populations of Bakiga, Rwandans and Baganda who mainly speak Runyankore dialect. The main economic activity is mixed farming and the main food crops grown include bananas, finger millet, beans, groundnuts, cowpeas, sweet potatoes, cassava, sorghum, maize, tomatoes, pineapples, passion fruits, sugar canes, mangoes and papaws. The population of the district is estimated to be 1,093,388. Females aged 15-49 years are estimated to make up 23% of the total population. Pregnant women are estimated to be 5.2% of the total population. The total fertility rate in Uganda is estimated at 6.9.

The study will be a randomised double-blind placebo-controlled trial with two arms. The researchers and the ANC staff will be blind to the HIV status of the mothers. However, mothers who choose to disclose their HIV status to the antenatal care staff are free to do so.

Difference in placental parasitaemia between HIV seropositive and HIV seronegative women was used to determine sample size. Using a power of 90% and a significance level of 5%, the sample size needed to detect a true difference in prevalence of maternal placental parasitaemia in the two study groups will be 104 women per group. However, to compensate for loss of follow-up, 30% will be added per group and this will give a total of 135 HIV seropositive women in each arm, giving a total of 270 HIV sero-positive mothers in the two study arms. Since HIV sero-prevalence in primigravidae attending antenatal care in the district is 10%, a minimum number of 1274 women would be required in each arm (total 2548).

Women will be enrolled in ANC clinics of three health units. All pregnant women, irrespective of parity, who consent to participate in the study will be enrolled.

Demographic and socio-economic characteristics will be recorded. History of fever and antimalarial drug use will also be recorded. Women will be randomly allocated to the SP + CQ (CQ 300 mg weekly) or SP + placebo group (IPT twice during pregnancy). All women will receive supplementation of 120mg elementary iron daily and 5mg folic acid weekly. IPT with SP will be started in the second trimester and a second dose in the third trimester. Women will be encouraged to deliver in health units and TBAs will be involved to follow-up of those who deliver in the villages. Health workers will liaise with TBAs to collect information and samples (birth weight and blood slides). The general health conditions of the mothers (including Hb, clinical malaria, body temperature, body weight, foetal heart sound, urine analysis) will be assessed throughout pregnancy. Clinical malaria cases will be treated according to national guidelines with CQ and SP. In case of treatment failure quinine will be given as second line treatment.

Inclusion and Exclusion Criteria:

All pregnant women presenting for ANC at the hospitals or health centres of study, irrespective of parity and consent to participate, will be enrolled in the study. Only women who consent to have an HIV test done and to be examined for viral load will be included. Women with at risk pregnancy, severe systemic disease or symptoms and signs of AIDS will be excluded from the study. Those women will be referred for further diagnosis and treatment at the nearest hospital.

Outcome Variables:

* maternal peripheral parasitaemia;
* placental parasitaemia;
* clinical malaria;
* maternal and infant Hb;
* birth weight;
* congenital parasitaemia;
* maternal HIV viral load at inclusion and before delivery.

Blood smears for parasitaemia will be made at enrolment, antenatal follow-up and delivery. Screening for HIV status will be done at enrolment and a confirmatory test done at the same time. Viral load will be assessed at enrolment and 36 weeks of gestation. At enrolment 5 ml of blood will be drawn for HIV screening, viral load and Hb measurement, and malaria parasitaemia assessment. Malaria parasites will be counted against 200 leukocytes and expressed as number of parasites/dl of blood assuming a standard leukocyte count of 8000/dl. The HIV status will be assessed using the existing Rapid Test used in the district for HIV screening.All women will receive pre- and post-screening counselling. Hb will be measured using a Haemo-Cue® portable photometer.

Compliance with the weekly CQ chemoprophylaxis will be controlled by giving the women a varying excess of tablets of CQ and placebo to take home and be requested to return the balance at each monthly visit. Health workers will administer the SP (DOT). The first dose of SP will be given at 14 - 24 weeks of gestation and the second dose will be given 28 - 32 weeks of gestation. Health workers will keep records of the gestational age.

Parasitaemia and Hb will be assessed at inclusion, at week 28 and at delivery. During monthly antenatal care visits women will be asked about illnesses that have occurred since their last visit and about any treatment taken. Routine ANC examinations will be undertaken. Malaria attacks will be recorded and women will be advised to come for treatment at the health units in case of any illness. Records will be kept by health care workers (laboratory staff, midwives, counsellors), TBAs and the PI. The District Director of Health Services (DDHS) will be an independent monitor for the research project.

Women presenting for delivery will be asked about recent malaria and other symptoms. Thick blood smears will be made from maternal peripheral blood, placental and umbilical cord blood. The newborn babies will be weighed with digital scales. At the onset of labour, the HIV sero-positive women will be treated with a single dose of 200mg Nevirapine and their newborn babies will also be treated with a single dose of 2mg/kg (or 0.6ml) Nevirapine within 72 hours after birth.

Health workers will be trained on how to use the Haemo-Cue® portable photometer and how to prepare thick blood slides. Since some women are likely to deliver in the villages, TBAs will be trained to weigh babies, prepare thick blood slides from the placenta for mothers that deliver in the villages. Blood samples for viral load if not taken before Nevirapine administration would lead to loss of follow-up of that woman.

For babies delivered in the villages, health workers will be informed as soon as possible to allow them to take the necessary measurements and also give the necessary assistance to the mothers and immunise the babies.

The qualitative component of the study will involve the use of FGD with pregnant women and mothers of neonates to assess their perceptions of the quality of maternity care services in their communities. In-depth interviews with health care providers providing maternity care services and drug sellers will be conducted to explore their perceptions on the quality of maternity care services and fever care seeking patterns of pregnant women in the study area. Illness narratives will be collected from pregnant women on their care seeking options and fever prevention strategies and practices during pregnancy.

Data Analysis:

Quantitative data will be analysed using SPSS and EPI INFO packages. Differences between proportions and means will be analysed using chi-square tests, ANOVA and Student t-tests. RR will be calculated. P value of < 0.05 will be considered significant.red to have significant difference or show statistical significance. Qualitative data will be coded for the themes of interest and emerging themes and a master sheet will be used to summarise the data from the different methods used to collect data. Ethnographic summaries, use of quotes and content analysis will be the methods used to analyse the qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* 14-24 weeks gestation
* Consent
* Presenting for ANC at study hospitals/centres
* Agree to have an HIV test and to be examined for viral load

Exclusion Criteria:

* Severe systemic disease
* AIDS-related disease
* At-risk pregnancy

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2548
Dates: Start 2003-08; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
maternal peripheral parasitaemia
placental parasitaemia
clinical malaria
maternal and infant Hb
birth weight
congenital parasitaemia
maternal HIV viral load at inclusion and before delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lucy N Korukiiko, MPH, Principal Investigator — Uganda AIDS Commission
Locations (1):
- Uganda AIDS Commission, Kampala, Kampala, Uganda

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- See also: DBL-Centre for Health Research and Development — http://www.dbl.life.ku.dk